CLINICAL TRIAL: NCT04237090
Title: Feasibility of a Randomized Controlled Clinical Trial Comparing the Use of Cetirizine to Replace Diphenhydramine in the Prevention of Reactions Related to Paclitaxel
Brief Title: Feasibility of a Clinical Trial Comparing the Use of Cetirizine to Replace Diphenhydramine in the Prevention of Reactions Related to Paclitaxel
Acronym: PREMED-F1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Matthieu Picard, Assitant clinical professor, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020-2110
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer; Lung Cancer; Ovarian Cancer; Oesophageal Cancer; Head Cancer Neck; Cervical Cancer; Endometrial Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Esophageal Neoplasms; Head and Neck Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — Diphenhydramine; Cetirizine; Lactose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Diphenhydramine + placebo (Active Comparator): Diphenhydramine 50 mg intravenous given in a 50 milliliters bag of sodium chloride 0.9 percent, with famotidine, 30 minutes before the paclitaxel infusion. 15 minutes infusion.
  Lactose tablet 100 mg per os given 30 minutes before the paclitaxel infusion.with a 180 milliliters glass of water.
  Interventions: Drug: Diphenhydramine; Drug: Lactose pill
- Cetirizine + placebo (Experimental): Cetirizine tablet 10 mg per os given 30 minutes before the paclitaxel infusion.with a 180 milliliters glass of water.
  1 milliliter of sodium chloride 0,9 percent intravenous given in a 50 milliliters bag of sodium chloride 0.9 percent, with famotidine, 30 minutes before the paclitaxel infusion. 15 minutes infusion.
  Interventions: Drug: Cetirizine; Drug: Sodium chloride 0.9%

INTERVENTIONS:
Drug: Diphenhydramine — Drug identification number : 02369567
  Other Names: Benadryl
  Arms: Diphenhydramine + placebo
Drug: Cetirizine — Drug identification number : 02231603
  Other Names: Reactine
  Arms: Cetirizine + placebo
Drug: Lactose pill — Natural product number : 00501190
  Arms: Diphenhydramine + placebo
Drug: Sodium chloride 0.9% — Drug identification number : 00037796
  Arms: Cetirizine + placebo

SUMMARY:
Explore the randomized, controlled, double-blind design targeted for the final clinical trial to assess the acceptability of interventions and clinical outcome measures and to provide data making it possible to estimate the parameters necessary for the preparation, modification or even abandonment of the final study.

DETAILED DESCRIPTION:
Paclitaxel is known to cause 30 to 40% of infusion-related reactions when no premedication is administered. It is agreed that all patients should receive premedication with dexamethasone, an H1 antagonist, such as diphenhydramine, and an H2 antagonist before the administration of paclitaxel. There are several cases where undesirable effects (eg. drowsiness, dry mouth, motor impatience) have been reported following the administration of this conventional premedication. Diphenhydramine is often accused because of its pharmacological properties.

A definitive, randomized, double-blind, non-inferiority study can assess whether cetirizine, a non-sedating H1 antagonist, can be used as an effective and safe alternative to diphenhydramine in the prevention of paclitaxel infusion-related reactions.

In the current proposed feasibility study, patients will be followed for the first two doses of paclitaxel. The goal is to explore the randomized, controlled, double-blind design targeted for the final clinical trial to assess the acceptability of interventions and clinical outcome measures and to provide data making it possible to estimate the parameters necessary for the preparation, modification or even abandonment of the final study.

ELIGIBILITY:
Inclusion Criteria:

* Receiving intravenous chemotherapy treatments at the Maisonneuve-Rosemont hospital outpatient oncology clinic
* Starting their first lifetime treatment with paclitaxel (alone or in combination with other anticancer agents).
* Capable of giving free and informed consent and who agrees to participate by signing the consent form
* Aged 18 and over
* Able to complete questionnaires

Exclusion Criteria:

* Does not understand French or English
* Taking chronic H1 antagonist orally
* Taking chronic systemic corticosteroids
* Contraindication or possible medical danger, such as a documented allergy or previous intolerance, related to the administration of cetirizine, diphenhydramine, placebo or any ingredient in their formulation
* Has received paclitaxel, docetaxel or paclitaxel nanoparticles linked to albumin in the past
* Receiving paclitaxel nanoparticles linked to albumin
* Severe renal impairment (Cockcroft-Gault <10 milliliters/minute)
* Pregnant or breastfeeding women
* Receiving paclitaxel under desensitization protocol
* Documented or reported dysphagia or other pathophysiological condition preventing a tablet from being swallowed whole
* Interactions preventing the full dose of oral cetirizine from being absorbed
* Participating in another clinical trial simultaneously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline of drowsiness on Stanford Sleepiness Scale 1 hour after the administration of diphenhydramine | 15 minutes before the administration of diphenhydramine. 1 hour after the administration of diphenhydramine.
  For treatment 1 and treatment 2
Change from baseline of drowsiness on Stanford Sleepiness Scale upon arrival at home | 15 minutes before the administration of diphenhydramine. Upon arrival at home.
  For treatment 1 and treatment 2
Change from baseline of drowsiness on Stanford Sleepiness Scale the morning after the administration of diphenhydramine | 15 minutes before the administration of diphenhydramine. Morning of day 2.
  For treatment 1 and treatment 2
Recruitment rate accomplished to recruit 24 participants for which a first dose of paclitaxel was administered between February and September 2020. | Through study completion, 8 months
  Number of participants per month recruited for which a first dose of paclitaxel was administered
Percentage of participants recruited, randomized and having received the first treatment of paclitaxel planned in the study between February and September 2020 following an assessment of their eligibility. | Through study completion, 8 months
  Number of participants recruited, randomized and having received the first treatment of paclitaxel planned in the study divided by the number of participants eligible to participate in the study

SECONDARY OUTCOMES:
Proportion of participants per group who required stopping the infusion and/or using rescue medication. | Day 1
  Stopping the infusion and using rescue medication defined by the medical choice of the attending physician. For treatment 1 and treatment 2.
Infusion-related reactions grade according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 classification | Day 1
  Grades will be determined using nurses notes. For treatment 1 and treatment 2

OTHER OUTCOMES:
Proportion of participants who completed the study | Through the course of the study, 8 months
  Number of participants who will have completed the study in each group divided by the number of participants recruited in each group
Reasons of loss to follow-up using a home-made questionnaire | Day 1
  For treatment 1 and treatment 2
Maintenance of the blind in participants using a home-made questionnaire | Day 1
  At the end of paclitaxel infusion of treatment 2
Maintenance of the blind in nurses using a home-made questionnaire | Day 1
  At the end of paclitaxel infusion of treatment 1 and 2
Side effects experienced by participants using a home-made questionnaire | Day 2
  Focus on drowsiness, dry mouth, eyes or nose, dizziness and restlessness/excitement. For treatment 1 and treatment 2.

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Picard, M.D., Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- CIUSSS de l'Est-de-l'île-de-Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiss RB, Donehower RC, Wiernik PH, Ohnuma T, Gralla RJ, Trump DL, Baker JR Jr, Van Echo DA, Von Hoff DD, Leyland-Jones B. Hypersensitivity reactions from taxol. J Clin Oncol. 1990 Jul;8(7):1263-8. doi: 10.1200/JCO.1990.8.7.1263. PMID 1972736
- [Background] Picard M, Castells MC. Re-visiting Hypersensitivity Reactions to Taxanes: A Comprehensive Review. Clin Rev Allergy Immunol. 2015 Oct;49(2):177-91. doi: 10.1007/s12016-014-8416-0. PMID 24740483
- [Background] Picard M. Management of Hypersensitivity Reactions to Taxanes. Immunol Allergy Clin North Am. 2017 Nov;37(4):679-693. doi: 10.1016/j.iac.2017.07.004. Epub 2017 Aug 18. PMID 28965634
- [Background] Durham CG, Thotakura D, Sager L, Foster J, Herrington JD. Cetirizine versus diphenhydramine in the prevention of chemotherapy-related hypersensitivity reactions. J Oncol Pharm Pract. 2019 Sep;25(6):1396-1401. doi: 10.1177/1078155218811505. Epub 2018 Nov 12. PMID 30419768
- [Background] Siderov J, Wendel N, Davis ID. Non-Sedating Antihistamines for Premedication in Ambulatory Oncology Patients. Journal of Pharmacy Practice and Research 2002; 32(2): 108-9.
- [Background] del Cuvillo A, Mullol J, Bartra J, Davila I, Jauregui I, Montoro J, Sastre J, Valero AL. Comparative pharmacology of the H1 antihistamines. J Investig Allergol Clin Immunol. 2006;16 Suppl 1:3-12. No abstract available. PMID 17357372
- [Background] Banerji A, Long AA, Camargo CA Jr. Diphenhydramine versus nonsedating antihistamines for acute allergic reactions: a literature review. Allergy Asthma Proc. 2007 Jul-Aug;28(4):418-26. doi: 10.2500/aap.2007.28.3015. PMID 17883909
- [Background] Berger MJ, Vargo C, Vincent M, Shaver K, Phillips G, Layman R, Macrae E, Mrozek E, Ramaswamy B, Wesolowski R, Shapiro CL, Lustberg MB. Stopping paclitaxel premedication after two doses in patients not experiencing a previous infusion hypersensitivity reaction. Support Care Cancer. 2015 Jul;23(7):2019-24. doi: 10.1007/s00520-014-2556-x. Epub 2014 Dec 18. PMID 25519756
- [Derived] Beaucage-Charron J, Gaudet L, Lamothe S, Pelletier C, Pepin AS, Roy V, Charpentier F, Lordkipanidze M, Projean D, Bouchard P, Picard M. A randomized double-blind feasibility study comparing cetirizine and diphenhydramine in the prevention of paclitaxel-associated infusion-related reactions: the PREMED-F1 study. Support Care Cancer. 2022 Apr;30(4):3389-3399. doi: 10.1007/s00520-021-06734-4. Epub 2022 Jan 8. PMID 34997314